## ClinicalTrials.gov ID NCT03990051

# Treatment Safety and Efficacy of Pro-ocular™ 1% for Chronic Ocular Graft Following Allogeneic HSCT

Sponsor: Glia, LLC

**Protocol** 

March 17, 2020

# TREATMENT FOR CHRONIC OCULAR GRAFT-VERSUS-HOST DISEASE - CLINICAL STUDY PROTOCOL -

| Protocol Title: Treatment safety and efficacy using Pro-ocular <sup>TM</sup> for chronic ocular graft versus host disease (GvHD) following allogeneic hematopoietic stem cell transplantation. | |
|---|---|
| Study Objective: | To evaluate the safety and efficacy of Pro-ocular <sup>TM</sup> 1% topical gel administered twice daily for 70 days in ameliorating symptoms and signs of chronic ocular GvHD. |
| Version / Date: | V 5.1 March 17, 2020 |
| <b>Protocol Number:</b> | oGvHD-1 |
| Study Phase: | 2 |
| Study Drug and Placebo: | Pro-ocular <sup>TM</sup> 1% topical gel (progesterone) and placebo |
| IND Number: | 143010 |
| Indication: | Reduce or eliminate ocular symptoms and signs of chronic ocular graft-versus-host disease |
| Study Site: | Massachusetts Eye and Ear Longwood<br>800 Huntington Avenue<br>Boston, MA 02115 |
| Principal Investigator: | Zhonghui Katie Luo, MD, PhD |
| Co-Investigators: | Edwin P. Alyea III, MD Joseph H. Antin, MD Philippe Armand, MD, PhD Corey S. Cutler, MDCM, MPH Mahasweta Gooptu, MD Vincent Trien-Vinh Ho, MD John Koreth, MBBS, DPhil Sarah Nikiforow, MD, PhD Rizwan Romee, MD Robert J. Soiffer, MD |
| Sponsor: | 134 Saint Botolph Street<br>Boston, MA 02115 |
| IRB: | Partners Human Research Committee |

## **Confidentiality Statement**

This protocol contains confidential, proprietary information of Glia, LLC. Further dissemination, distribution or copying of this protocol or its contents is strictly prohibited

#### Approved:

Zhonghui Katie Luo, MD, PhD, Principal Investigator Robert J. Soiffer, MD, Co-Investigator Wei-wei Chang, PhD, GLIA LLC Kenneth Sawyer, JD, GLIA, LLC

#### **CONTACT INFORMATION FOR THE STUDY**

| Principal Investigator: | Zhonghui Katie Luo, MD, PhD |
|---|---|
| | MEE Longwood |
| | 800 Huntington Avenue |
| | Boston, MA 02115 |
| | Email: Zhonghui_Luo@MEEI.Harvard.edu |
| Administrative Contact: | Patricia Li |
| | Tel. 617-936-6092 (7:30 am – 3:30 pm) |
| | Partners Human Research Committee |
| IRB: | 399 Revolution Drive |
| | Suite # 710 |
| | Somerville MA, 02145 |
| | 857-282-1900 |
| <b>Sponsor Contact:</b> | Wei-wei Chang, PhD |
| | Direct: 617-794-8922; email <a href="mailto:chang@gliacell.com">chang@gliacell.com</a> |
| | Kenneth Sawyer, JD |
| | Direct: 201-621-1036; email sawyer@gliacell.com |
| | Glia, LLC |
| | 134 Saint Botolph Street |
| | Boston, MA 02115 |
| | Tel: 617-859-0800 |
| | Fax: 617-859-0818 |

## **SYNOPSIS**

| Protocol Title: | Treatment safety and efficacy using Pro-ocular <sup>TM</sup> for chronic ocular graft versus host disease (GvHD) following allogeneic hematopoietic stem cell transplantation |
|---|---|
| Version / Date: | V 5.1 March 17, 2020 |
| Protocol Number: | oGvHD-1 |
| Study Phase: | 2 |
| Study Drug and Placebo: | Pro-ocular <sup>TM</sup> 1% topical gel (progesterone USP) and placebo |
| IND Number: | 143010 |
| Indication: | Reduce or eliminate ocular symptoms and signs of chronic ocular graft-versus-host disease |
| Study Objective: | To evaluate the safety and efficacy of Pro-ocular™ 1% topical gel administered twice daily for 70 days in ameliorating symptoms and signs of chronic ocular GvHD. |
| Design Structure: | Single center, randomized, parallel, double-masked, placebo-controlled study |
| Institutional Review Board: | Partners Human Research Committee |
| Duration: Dosage/Dose Regimen: | 10-week treatment period (active and placebo) 6-week crossover period (placebo to active) open label phase long term phase to extend the entire treatment period for 27 months Approximately 0.07 g Pro-ocular <sup>TM</sup> 1% topical gel applied and massaged into the forehead skin twice daily, |
| Route of Administration: | morning and before bedtime. Area of Application |
| Visit Schedule, Double-Masked<br>Phase: | <ul> <li>5 visits over 70 days including:</li> <li>Visit 1, Screening (Day -14 to -1)</li> <li>Visit 2, Baseline and 1<sup>st</sup> drug application</li> <li>Visit 3, 2-week follow-up (Day 14 ± 2)</li> <li>Visit 4, 6-week follow-up (Day 42 ± 3)</li> <li>Visit 5, 10-week follow-up (Day 70 ± 3)</li> </ul> |
| Crossover Phase for Subjects on Placebo: | Subjects in placebo group will receive Pro-ocular 1% topical gel for twice daily administration for over 6 weeks starting at Visit 5: |

| | <ul> <li>Visit 6, 13-week follow-up (3 weeks on active drug), placebo cross-over subjects only</li> <li>Visit 7, 16-week follow-up (6 weeks on active drug), placebo cross-over subjects only</li> </ul> |
|---|---|
| Long Term Follow Up for<br>Subjects in Open Label Phase<br>(for Eligible & Interested<br>Subjects) | Drug will be supplied after the study period for a total of 27 months' treatment period beginning with Visit 2, with safety monitoring and reporting by the PI and co-investigators under protocol during clinic: Visit 8, 66 ± 6 weeks (15 months) Visit 9, 117 ± 6 weeks (27 months) |
| Measures Taken to Reduce Bias: | Randomized treatment assignment; double-masked parallel study design, 2:1, study drug: placebo, 22 subjects:11 subjects |
| Number of Subjects: | 33 patients diagnosed with chronic ocular GvHD in at least one eye, not wearing scleral or contact lens for at least one month in any eye prior to screening |
| Number of Study Sites: | 1 |
| Inclusion Criteria: | <ol> <li>Male or female of any race, at least 18 years of age at Visit 1 Screening.</li> <li>Has the diagnosis of chronic ocular GvHD.</li> <li>Has the NIH Consensus Eye Score of at least 2.</li> <li>On the GLIA Ocular Surface Disease Symptoms Questionnaire at Screening, has ocular discomfort at a severity score of moderate or more, and at least one other symptom at a severity of moderate or more.</li> <li>One or more signs from the list of chronic ocular GvHD signs below.</li> <li>Has provided verbal and written informed consent.</li> <li>Be able and willing to follow oral and written instructions, including participation in all study assessments and visits.</li> </ol> |
| Exclusion Criteria: | <ol> <li>Wearing scleral lens within the last month, or those who plan to start wearing scleral lens during the study.</li> <li>Anticipate major changes in systemic GvHD management during study period.</li> <li>Comorbidity with other severe or chronic eye conditions that in the judgment of the investigator will interfere with study assessments, such as but not limited to retinal detachment, recent ocular surgery, Bell's palsy, active trigeminal neuritis or neuralgia.</li> </ol> |

- 4. Anticipate change of vision correction or anticipate any ocular procedure during study period.
  - 5. A woman who is pregnant, nursing an infant, or planning a pregnancy.
- 6. A woman of childbearing potential who has a positive urine pregnancy test at Visit 1, or who does not use an adequate method of birth control throughout the study period.
- 7. Has a known adverse reaction and/or sensitivity to the study drug or its components.
- 8. Unwilling to cease the use of sunscreen on the forehead or eye area.
- 9. Intraocular pressure >22 mm Hg at screening visit with or without ongoing glaucoma treatment.
- 10. Currently enrolled in an investigational drug or device study for ocular GvHD.

#### **Evaluation Criteria:**

#### **Efficacy Measures:**

Glia Ocular Surface Disease Symptoms Questionnaire, Clinic and Daily Diary

- Ocular discomfort
- Dryness
- Grittiness
- Burning
- Stinging
- Foreign body sensation
- Ocular pain
- Conjunctival redness
- Itching
- Photophobia
- Mucus discharge
- Blurred or cloudy vision
- Air flow sensitivity
- Lid redness
- Lid sticking

Daily use of eye drops (Restasis®, Xiidra®, artificial tears and/or gels, autologous tears (# times administered per wake-time hours and sleep-time hours)

SANDE – Symptom Assessment iN Dry Eye

Ouestionnaire

National Institutes of Health Eye Score Chronic ocular GvHD Signs (Ophthalmologist examination at each visit)

- TearScan examination: Tear film, lid margins, and meibum expression

| | <del>_</del> |
|---|---|
| | <ul> <li>Visual acuity with current correction.</li> <li>Slit lamp without staining: Lids (lid margin erythema, edema, ulceration, notches, entropion/ectropion, trichiasis/madarosis, floppy eyelids, hordeolum); Conjunctiva (hyperemia, cicatricial changes, pseudomembranes, chalasis); Cornea (edema, ulcers, filamentous keratitis, thinning, corneal neovascularization, scars, conjunctival epithelium invasion, limbal thickening).</li> <li>Corneal and conjunctival fluorescein staining Non-Ocular GvHD Signs (recorded by patient and physician):</li> </ul> |
| | - Systemic assessment by BMT physician such as |
| | dry mouth |
| Safety Measures: | <ul> <li>Adverse events</li> <li>Visual acuity</li> <li>Slit lamp biomicroscopy</li> <li>Undilated fundoscopy examination</li> <li>Intraocular pressure</li> <li>Systemic assessment by BMT physician at Dana<br/>Farber Cancer Institute</li> </ul> |
| Laboratory Tests Routine and<br>Afor Assessment of HPA<br>(hypothalamic-pituitary-<br>adrenal axis) Function | Tests to be run at Visits 1, 4, 5, 7, 8 and 9: Standard panel to include CBC with differential, metabolic panel, tacrolimus/sirolimus levels, Vitamin D Total 25-hydroxy (D2 and D3), T4 (T total and free), T3, ACTH, TSH, DHEA-S, estradiol, FSH, LH, progesterone, testosterone (total and free). |

# TREATMENT FOR CHRONIC OCULAR GRAFT-VERSUS-HOST DISEASE CLINICAL STUDY PROTOCOL

## **Table of Contents**

| SYN | OPSIS | 3 |
|---|---|---|
| List | of Abbreviations | 8 |
| TRE | ATMENT FOR CHRONIC OCULAR GRAFT-VERSUS-HOST DISEASE - CLINICAL STUDY PROTOCOL | <u>S</u> |
| l. | BACKGROUND AND SIGNIFICANCE | <u>S</u> |
| II. | SPECIFIC AIMS | 10 |
| III. | SUBJECT SELECTION | 10 |
| IV. | SUBJECT ENROLLMENT | 12 |
| V. | STUDY PROCEDURES | 12 |
| VI. | BIOSTATISTICAL ANALYSIS | 18 |
| VII. | RISKS AND DISCOMFORTS | 19 |
| VIII. | POTENTIAL BENEFITS | 19 |
| IX. | MONITORING AND QUALITY ASSURANCE | 20 |
| X. | REFERENCES | 21 |
| APP | PENDICES | 26 |
| SCH | IEDULE OF VISITS AND ASSESSMENTS | 27 |
| Visit | ts 1-7 | 27 |
| SCH | EDULE OF VISITS AND ASSESSMENTS | 28 |
| Visit | ts 8-10 Long Term Open Label | 28 |

#### **List of Abbreviations**

ADL Activities of daily living

AE Adverse event BID Twice a day

BMT Bone marrow transplantation

CN V Cranial Nerve Five CN VII Cranial Nerve Seven CS Clinically significant

CTCAE Common Terminology Criteria for Adverse Events

CV Curriculum vitae

FDA Food and Drug Administration

g gram

GvHD Graft-versus-host disease

HSCT Hematopoietic stem cell transplantation

ICF Informed consent form

IND Investigational new drug application

IOP Intraocular pressure
IRB Institutional review board

ITT Intent to treat kg kilogram

LOCF Last observation carried forward

MedDRA Medical Dictionary for Regulatory Activities

 $\begin{array}{ccc} mg & milligram \\ \mu g & microgram \\ mL & milliliter \\ \mu L & microliter \\ mm & millimeter \\ \mu m & micrometer \\ \end{array}$ 

mmHg millimeters of mercury NCS Not clinically significant

nd not done OD Right eye

oGvHD Ocular graft-versus-host disease

OS Left eye OU Both eyes

SAE Serious adverse event SAP Statistical analysis plan SD Standard deviation

USP United States Pharmacopeia

VA Visual acuity

## TREATMENT FOR CHRONIC OCULAR GRAFT-VERSUS-HOST DISEASE - CLINICAL STUDY PROTOCOL

#### I. BACKGROUND AND SIGNIFICANCE

#### a. Historical background

Pro-Ocular™ topical gel has been studied in controlled clinical studies for dry eye, ocular discomfort and in compassionate use since 2013. Each metered dose of Pro-Ocular 1% will be about 0.07 g containing about 0.7 mg progesterone. One skin penetration study showed that less than 5% of the applied dose was able to cross the outer skin layer or stratum corneum.

#### b. Scientific evidence

The animal study done by Ian Meng et.al has just been published on Investigative Ophthalmology & Vision Science 2019; 60 (1706-1713). The study has shown that Progesterone 1% gel application to the forehead, but not the contralateral cheek of the rats, decreased pain sensation from capsaicin and hypertonic saline application. Local anesthesia of the forehead skin blocks the response. The work has indicated that the mechanism of action is not via systemic absorption; and a local neuro-pathway is likely activated to alter corneal nociception, likely via the cranial nerve V1 branch.

c. Previous pre-clinical or clinical studies leading up to, and supporting the proposed research

A product with a similar formulation, PG101 1% topical gel, was given to 24 subjects in a completed clinical trial for dry eyes under US IND 119774. A second group consisting of 24 subjects received PG101 0.25%. No drug related serious adverse events were reported. Adverse events with potential relationship to the topical gels in the completed study are approximately equal in placebo and treatment groups. The product demonstrated efficacy in multiple symptoms of dry eye disease such as ocular discomfort, dryness, and grittiness in both active arms as well as central corneal staining in the 1% active arm.

A study under US IND 123266 for ocular discomfort in glaucoma patients involving 0.5% topical gel enrolled approximately 40 subjects with no potential drug related serious adverse events reports. The study has not been unblinded for efficacy analysis.

Since late 2015 Pro-Ocular<sup>TM</sup> topical gel has been used by a total of 15 chronic ocular GvHD patients who had been suffering extreme ocular discomfort, with almost all encountering intractable ocular pain despite treatment with all available ocular drugs and devices such as BostonSight PROSE (prosthetic replacement of the ocular surface ecosystem). For most patients relief in symptoms began with the first application, and greater relief ensued with additional use. Symptomatic improvements to various extend were achieved by all patients after several weeks. For those wearing scleral lens, daily discomfort during wear and accumulation of debris behind the lens was reduced or eliminated.

Topical gels of both concentrations have been prescribed and dispensed through an authorized compounding pharmacy to additional patients under care of ophthalmologists. The prescribing physicians reported no serious treatment-related adverse events.

The same active ingredient, progesterone USP, occurs naturally in the human body, male and female, and can reach levels as high as 100-200 ng/mL during late pregnancy. It is administered

at high doses in marketed FDA-approved products orally (200-400 mg/day), vaginally (300-800 mg/day), intramuscularly (up to 10 mg/day), and topically in marketed supplements (up to 80 mg/day). Both progesterone prescription products and marketed supplements are used chronically.

Progesterone is also found in foods such as eggs, dairy, yams, beans and dark green leafy vegetables.

c. Rationale behind the proposed research, and potential benefits to patients and/or society

A controlled study is necessary to verify findings in isolated patients, and is required for product to be approved by the Food and Drug Administration in order that the product can be made available to other patients. Currently available ophthalmic solutions and suspensions, drugs and devices have not been effective in alleviating the suffering of the ocular GvHD patients. Thus this is an unmet need that Pro-Ocular<sup>TM</sup> topical gel can fulfill.

Potential benefits: Decrease or cessation of adverse ocular symptoms and signs to regain quality of life, and prevention of ocular disease progression.

#### II. SPECIFIC AIMS

To evaluate the safety and efficacy of Pro-Ocular™ 1% topical gel administered twice daily for 70 days in ameliorating symptoms and signs of chronic ocular GvHD.

#### III. SUBJECT SELECTION

The plan is to screen 42 patients in order to achieve a study completion of 33 patients, 2:1 active drug:placebo. Subjects at least 18 years of age with a diagnosis of chronic ocular GvHD and fulfilling certain inclusion and exclusion criteria will be eligible. We anticipate that Dr. Luo, Principal Investigator, Ophthalmologist at MEE Longwood will have a sufficient number of eligible patients to enable enrollment from one site.

The inclusion and exclusion criteria are as follows:

| | 1. | 1. Male or female of any race, at least 18 years of age at |
|---|---|---|
| | | Visit 1 Screening. |
| | 2. | Has the diagnosis of chronic ocular GvHD. |
| | 3. | Has the NIH Consensus Eye Score of at least 2. |
| | 4. | On the GLIA Ocular Surface Disease Symptoms |
| Inclusion Criteria: | | Questionnaire at Screening, has ocular discomfort at a |
| | | severity score of moderate or more, and at least one |
| | | other symptom at a severity of moderate or more. |
| | 5. | One or more signs from the list of chronic ocular |
| | | GvHD signs below. |
| | 6. | Has provided verbal and written informed consent. |

| | 7. Be able and willing to follow oral and written instructions, including participation in all study |
|---|---|
| | assessments and visits. |
| Exclusion Criteria: | , 01 |
| | study for ocular GvHD. |

The definition of scoring from the NIH Consensus for ocular GvHD is as follows:

NIH Consensus: 2014 Diagnosis and Staging Working Group

| | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| EYES | No symptoms | Mild dry eye | Moderate dry eye | Severe dry eye |
| | | symptoms not | symptoms partially | symptoms significantly |
| Keratoconjunctivitis | | affecting ADL | affecting ADL | affecting ADL (special |
| sicca (KCS) confirmed | | (requirement of | (requiring lubricant | eyeware to relieve pain) |
| by ophthalmologist: | | lubricant eye | eye drops $> 3$ x per | OR unable to work |
| Yes | | drops $\leq 3 \times per$ | day or punctal | because of ocular |
| No | | day) | plugs), | symptoms OR loss of |
| Not examined | | | WITHOUT new | vision due to KCS |
| | | | vision impairment | |
| | | | due to KCS | |

#### IV. SUBJECT ENROLLMENT

#### a. Methods of enrollment

Dr. Luo will review the qualifications of her active chronic ocular GvHD patients to determine eligibility, and query the eligible patients via a phone call by Dr. Luo herself as to their interest in participation.

#### b. Procedures for obtaining informed consent

An informed consent form will be provided for eligible patients to review. Dr. Luo herself will obtain the informed consent with each subject.

#### c. Treatment assignment, and randomization

Randomized double-masked parallel treatment assignment will be made using a block design at the ratio of 2:1, study drug:placebo, 22:11.

#### V. STUDY PROCEDURES

The sequence of procedures at each clinic visit is as follows:

| Visit 1 (Day -14 to -1) |
|-----------------------------------------|
| Screening |
| Ophthalmology assessment |
| Informed consent by investigator |
| 2-digit subject ID number |
| GLIA Ocular GvHD symptoms questionnaire |
| SANDE symptoms questionnaire |
| NIH Ocular GvHD score |
| Visual acuity with current correction |
| Slit-lamp biomicroscopy |
| Undilated fundoscopy exam |
| Corneal and conjunctival staining |
| Intraocular pressure |
| Urine pregnancy testing (as needed) |
| Inclusion/Exclusion criteria |

Screening Pass or Fail by investigator
Subject assigned 3-digit randomization code
Review medical records for medical & ocular history
Review prior and current medications
Demographics

#### BMT (DFCI) physician systemic evaluation

History

Physical

Concomitant medications
Laboratory tests, standard & endocrine panel
GvHD assessment

1

#### Visit 2 (Day 1)

#### **Baseline & First Drug Application**

Medical/ocular update
Medication update
Facial photo

1 minute video of face and eyes (+ blink interval)
TearScan examination
GLIA Ocular GvHD symptoms questionnaire
Dispense study drug by investigator
STUDY DRUG APPLICATION by investigator
30-90 minutes' wait from application

1 minute video of face and eyes (+ blink interval)
TearScan examination

Adverse event query
GLIA Ocular GvHD symptoms questionnaire
Dispense daily diary and ocular medication log



#### Visit 3 (Day 14 ± 2), 2 weeks' treatment

Medical and medication update
Diary and ocular medication log collection & compliance
Drug collection & accountability

1 minute video of face and eyes (+ blink interval)

TearScan examination
Adverse event query
SANDE symptoms questionnaire
GLIA Ocular GvHD symptoms questionnaire
Slit-lamp biomicroscopy
Corneal and conjunctival staining
Study drug, daily diary and ocular medication log dispensed



#### Visit 4 (Day 42 ± 3), 6 weeks' treatment

#### **Ophthalmology assessment**

Medical and medication update
Diary and ocular medication log collection & compliance

Drug collection & accountability

1 minute video of face and eyes (+ blink interval)

TearScan examination

Adverse event query

SANDE symptoms questionnaire

GLIA Ocular GvHD symptoms questionnaire

Slit-lamp biomicroscopy

Corneal and conjunctival staining

Study drug, daily diary and ocular medication log dispensed

#### BMT(DFCI) physician systemic evaluation

Standard lab tests, GvHD assessment



#### Visit 5 (Day 70 ± 3), 10 weeks' treatment

#### **Ophthalmology assessment**

Visual acuity

Medical and medication update
Diary and ocular medication collection & compliance
Drug collection & accountability
Urine pregnancy test if applicable
Facial photo

1 minute video of face and eyes (+ blink interval)

TearScan examination

Adverse event query

SANDE symptoms questionnaire

GLIA Ocular GvHD symptoms questionnaire

Slit-lamp biomicroscopy

Undilated fundoscopy exam

Corneal and conjunctival staining

NIH Ocular GvHD score

Intraocular pressure

Urine pregnancy test

End of study phase

Reconfirm drug dispensing for Open label Phase
Dispense diary, ocular medication log and drug to Placebo

#### BMT (DFCI) physician systemic evaluation

Concomitant medications
Laboratory tests, standard & endocrine panel
GvHD assessment



### Visit 6, 13 weeks for Placebo group only

Medical and medication update
Diary and ocular medication log collection & compliance
Drug collection & accountability

1 minute video of face and eyes (+ blink interval)

TearScan examination
Adverse event query

SANDE symptoms questionnaire

GLIA Ocular GvHD symptoms questionnaire Slit-lamp biomicroscopy Corneal and conjunctival staining



#### Visit 7, 16 weeks for Placebo group only

Facial photo

Medical and medication update
Diary and ocular medication log collection & compliance

Drug collection & accountability

1 minute video of face and eyes (+ blink interval)

TearScan examination

Adverse event query

SANDE symptoms questionnaire

GLIA Ocular GvHD symptoms questionnaire

NIH Ocular GvHD Score<sup>1</sup>

Slit-lamp biomicroscopy

Corneal and conjunctival staining

Intraocular pressure

#### BMT (DFCI) physician systemic evaluation

Concomitant medications
Laboratory tests, standard & endocrine panel

GvHD assessment

# Long Term Follow Up for Subjects in Open Label Phase (for Eligible & Interested Subjects) Visit 8, 66 weeks ± 6 weeks (15 months)

Facial photo

1 minute video of face and eyes (+ blink interval)

TearScan examination

Adverse event query

SANDE symptoms questionnaire

GLIA Ocular GvHD symptoms questionnaire

NIH Ocular GvHD Score

Slit-lamp biomicroscopy

Visual Acuity

Undilated fundoscopy exam

Corneal and conjunctival staining

Intraocular pressure

#### BMT (DFCI) physician systemic evaluation

Concomitant medications

Laboratory tests

**GvHD** assessment

Long Term Follow Up for Subjects in Open Label Phase (for Eligible & Interested Subjects)

Visit 9, 117 ± 6 weeks (27 months)

Facial photo

-

<sup>&</sup>lt;sup>1</sup> Added as protocol deviation to original protocol v4.

1 minute video of face and eyes (+ blink interval)

TearScan examination

Adverse event query

SANDE symptoms questionnaire

GLIA Ocular GvHD symptoms questionnaire

NIH Ocular GvHD Score

Slit-lamp biomicroscopy

Visual Acuity

Undilated fundoscopy exam

Corneal and conjunctival staining

Intraocular pressure

#### BMT (DFCI) physician systemic evaluation

Concomitant medications
Laboratory tests, standard and relevant panel
GvHD assessment

## The evaluation criteria are as follows:

| Efficacy Massures | Clia Ogular CyllD Symptoma Ovactionnaira |
|---|---|
| <b>Efficacy Measures:</b> | Glia Ocular GvHD Symptoms Questionnaire |
| | Clinic Daily Diary |
| | - Ocular discomfort |
| | - Dryness |
| | - Grittiness |
| | - Burning |
| | - Stinging |
| | <ul> <li>Foreign body sensation</li> </ul> |
| | - Ocular pain |
| | - Conjunctival redness |
| | - Itching |
| | - Photophobia |
| | - Mucus discharge |
| | - Blurred or cloudy vision |
| | - Air flow sensitivity |
| | - Lid redness |
| | - Lid sticking |
| | Use of eye drops (Restasis®, Xiidra®, artificial tears and/or |
| | gels, autologous tears, # times administered per wake-time |
| | hours and sleep-time hours) |
| | SANDE – Symptom Assessment iN Dry Eye Questionnaire |
| | National Institutes of Health Eye Score |
| | Ocular GvHD Signs (physician examination at each visit) |
| | - TearScan examination: Tear film, lid margins, and |
| | meibum expression. |
| | - Visual acuity with current correction. |
| | - Slit lamp without staining: Lids (lid margin erythema, |
| | edema, ulceration, notches, entropion/ ectropion, |
| | trichiasis/madarosis, floppy eyelids, hordeolum); |
| | Conjunctiva (hyperemia, cicatricial changes, |
| | pseudomembranes, chalasis); Cornea (edema, ulcers, |
| | filamentous keratitis, thinning, corneal |
| | neovascularization, scars, conjunctivial epithelium |
| | invasion, limbal thickening). |
| | - Corneal and conjunctival fluorescein staining |
| | Non-Ocular GvHD Signs (recorded by patient and physician): |
| | - Systemic assessment by BMT physician such as dry |
| | mouth |
| | -140 9941 |
| | - Adverse events |
| | - Visual acuity |
| | - Slit lamp biomicroscopy |
| Safety Measures: | - Undilated fundoscopy examination |
| | - Intraocular pressure |
| | - Systemic assessment by BMT physician at Dana Farber |
| | Cancer Institute |
| Laboratory Tests | Tests to be run at Visits 1, 4, 5, 7, 8, and 9: CBC with |
| Routine and for | differential, metabolic panel, tacrolimus/sirolimus levels, |
| Toutine and for | annotation, memorite paner, actionnias/sitonnias tevels, |

| Assessment of HPA | Vitamin D Total 25-hydroxy (D2 and D3), T4 (Total and free), |
|---|---|
| (hypothalamic- | T3, ACTH, TSH, DHEA-S, estradiol, FSH, LH, progesterone, |
| pituitary-adrenal axis) | testosterone (total and free). |
| Function | |

Laboratory tests will be performed at the Dana Farber Cancer Institute (DFCI) and the Brigham Research Assay Core, Brigham and Women's Hospital. As DFCI patients study subject will continue to be followed at DFCI by the MD that referred them to Mass Eye and Ear. In addition to their standard of care examinations the study subjects will undergo additional laboratory testing including:

- CBC with differential
- Metabolic panel
- Tacrolimus/sirolimus levels
- Vitamin D Total 25-hydroxy (D2 and D3)
- T4 (Total and free)
- T3
- ACTH
- TSH.
- DHEA-S
- Estradiol
- FSH
- LH
- Progesterone
- Testosterone (total and free).

These DFCI physicians will be co-investigators in the study and will review the laboratory tests outcomes to ensure the safety of the subjects.

A selection of the key questionnaires and examination procedures specific to oGvHD are shown in the **Appendix**.

#### VI. BIOSTATISTICAL ANALYSIS

#### **Analysis Populations:**

#### Intent-to-Treat Population

The intent-to-treat (ITT) population includes all randomized subjects. The efficacy analyses will be performed on the ITT population with Last Observation Carried Forward (LOCF) method for missing values. The efficacy variables may also be analyzed utilizing the ITT population with observed data only (i.e. without LOCF) to assess sensitivity.

#### Per-Protocol Population

The per protocol (PP) population excludes subjects with significant protocol deviations and excludes any incomplete subject data. Protocol deviations will be assessed by the clinical team, prior to database lock. Efficacy analyses will be performed on the PP population with observed data only.

#### Sample Size

33 subjects.

#### **Efficacy Analyses**

The continuous and ordinal efficacy variables collected at each visit (and time point, where relevant) will be summarized with number of observations (n), mean, standard deviation, median, minimum and maximum. Statistical inference testing will be conducted and the results will be utilized as additional descriptors of the data. Two-sample *t*-tests will be employed for continuous variables. Two-sample t-tests, Wilcoxon rank sum tests and analysis of covariance (ANCOVA) models adjusting for baseline will be employed for ordinal variables. For the ANCOVA models, treatment will be compared to the placebo. Pearson's chi-square or Fisher's exact tests (in the case of expected counts less than 5) will be employed for qualitative variables. Where appropriate, the change from baseline for each parameter will also be summarized using descriptive statistics.

The individual symptoms collected in the diary will be analyzed including all data across the 70-day treatment period, testing for a treatment effect using a generalized linear model that accounts for repeated measures with an unstructured correlation structure, including terms for diary day and the treatment-by-day interaction.

#### VII. RISKS AND DISCOMFORTS

Based on the clinical use of the drug within and outside of controlled studies, there are no known risks. The amount of the active progesterone is several hundred-fold lower than the current injectable, topical, and oral forms. Skin penetration studies by Sponsor using the Franz cell has shown that less than 5% of progesterone passes through the top layer of the skin (stratum corneum).

Use of other ocular medications can continue, concurrent with use of Pro-ocular.

#### VIII. POTENTIAL BENEFITS

a. Potential benefits to participating individuals

The potential benefits to participating individuals are reduction or elimination of ocular discomfort, especially the extreme pain experienced by many ocular GvHD patients, and ocular tissue damage repair, potentially preventing progression to when surgical procedures may be required.

Another potential benefit is the reduction of use of artificial tears and other eye drops that only provide temporary relief.

There is potential improvement of the overall quality of life, and enabling the return to normal daily living, sleep, work, and other activities.

b. Potential benefits to society

The study is expected to prove that the study drug fulfills an unmet need for ocular GvHD treatment.

#### IX. MONITORING AND QUALITY ASSURANCE

a. Independent monitoring of source data

The sponsor intends to provide independent monitoring to ensure all data are collected, and entered into a database accurately.

#### b. Safety monitoring

A Safety Management Plan is provided to clinical management personnel. A 24-hour telephone physician safety monitor line will be provided for the subjects to call.

#### c. Outcomes monitoring

Data will be analyzed by a third-party statistical group.

#### d. Adverse event reporting guidelines

All adverse events will be collected, whether potentially related or unrelated to study drug use. The adverse events will be categorized according to the latest version of MedDRA (Medical Dictionary for Regulatory Activities) using Common Terminology Criteria (CTCAE). The Safety Management Plan provides guidance for what is considered a serious adverse event, the forms to be completed in such cases, and when a serious adverse event needs to be reported to the FDA.

## X. REFERENCES

## **Ocular Findings in Chronic GvHD**

| Reference | Ocular Changes Chronic GvHD |
|---|---|
| Amparo F et al. Corneal fluorescein staining and ocular symptoms but not Schirmer test are useful as indicators of response to treatment in chronic ocular GVHD. Ocul Surf. 2018 May 12. pii: S1542-0124(18)30040-5. | Corneal fluorescein staining and symptoms better indicators than Schirmer scores |
| Anderson NG, Regillo C Ocular manifestations of graft versus host disease. Curr Opin Ophthalmol. 2004 Dec;15(6):503-7. | "Ocular findings include keratoconjunctivitis sicca, pseudomembranous conjunctivitis, corneal ulceration and perforation, and microvascular retinopathy." |
| Berchicci L et al. Ocular chronic graft-versus-host disease after allogeneic hematopoietic stem cell transplantation in an Italian referral center. Ocul Surf. 2018 Jul;16(3):314-321. | More than 50% developed chronic ocular GVHD after allogeneic HSCT. Meibomian gland dysfunction, conjunctival hyperemia, and conjunctival fibrosis were major findings. |
| Blecha C et al. Verification of the new grading scale for ocular chronic graft-versus-host disease developed by the German-Austrian-Swiss consensus conference on chronic GVHD. Ann Hematol. 2016 Feb;95(3):493-9. | "85% of patients suffered from functional impairment due to ocular cGVHD." Ocular tissue involved: Lacrimal glad dysfunction 100% Lids 89% Conjunctiva 96% Cornea 76% |
| Blecha C et al. Retinal Involvement in a Patient with Cerebral Manifestation of Chronic Graft-Versus-Host-Disease. Oncol Res Treat. 2015;38(10):532-4. | "2 years later, she complained of right-sided blurred vision and floaters; both eyes showed whitish circumscribed retinal infiltrations, cellular infiltration of the vitreous and mild bilateral optic disc edema. Oncological and neurological work-up ruled out infectious diseases and other GvHD manifestations. Symptoms and signs resolved under continued systemic IS, leaving pigmented retinal scars." |
| Busin M, Giannaccare G, Sapigni L, Testoni N, Leon P, Versura P, Campos E. Conjunctival and Limbal Transplantation From the Same Living-Related Bone Marrow Donor to Patients With Severe Ocular Graft-vs-Host Disease. JAMA Ophthalmol. 2017 Oct 1;135(10):1123-1125. | "To date, no treatment has proven to be effective for severe ocular graft-vs-host disease (GVHD) after allogenic hematopoietic stem cell transplantation that leads to conjunctivalization and keratinization of the cornea through damage of conjunctival goblet cells and limbal epithelial stem cells (LESCs). We report the outcomes of chimerism induced by transplantation from the same living-related bone marrow donor of conjunctiva and LESCs in 4 eyes of 2 patients with severe ocular GVHD." |
| Claes K, Kestelyn P Ocular manifestations of graft versus host disease following bone marrow transplantation. Bull Soc Belge Ophtalmol. 2000;(277):21-6. | "The ocular manifestations of Graft Versus Host Disease (GVHD) include keratoconjunctivitis sicca, cicatricial lagophthalmos, sterile conjunctivitis, corneal epithelial defects, corneal ulceration and melting." |

| Reference | Ocular Changes Chronic GvHD |
|---|---|
| Curtis LM et al. Predictive models for ocular chronic graft-versus-host disease diagnosis and disease activity in transplant clinical practice. Haematologica. 2015 Sep;100(9):1228-36. | Significant findings in ocular cGvHD patients: Visual acuity deficits and vision difficulty Corneal staining Meibomian glands plugged Lid margin swelling Lid margin erythema Lid margin tear film debris Conjunctival injection [hyperemia → pseudomembranous conjunctivitis] Conjuntival chemosis [swelling] Dry eye (Schirmer test and tear film breakup time not as valuable as indicators.) |
| Dierich-Ntoukas T<br>[Clinical Signs of Ocular Graft-versus-Host Disease]. Klin<br>Monbl Augenheilkd. 2015 May;232(5):647-51. | "It is not only associated with reduced quality of life because of dry eye symptoms but can also impair visual acuity and lead to blindness due to corneal complications. Patients with ocular GvHD are often resistant to therapy because of the severe dry eye disease and persistent inflammatory activity." |
| Eberwein P et al<br>[Patient-Centred Care of Ocular Graft-vs-Host Disease in<br>Germany]. Klin Monbl Augenheilkd. 2015<br>May;232(5):664-8. | "Ocular GvHD is a severe complication following allogenic blood stem cell transplantation leading to massive reduction in quality of life and ocular pathologies including corneal perforation." |
| Gama I et al. Chronic Ocular Graft vs Host Disease as a Serious Complication of Allogeneic Hematopoietic Stem Cell Transplantation: Case Report. Transplant Proc. 2015 May;47(4):1059-62. | "Bilateral corneal ulcers and ocular perforation, although not frequent, can occur in most extreme cases." |
| Giannaccare G et al. Ocular surface analysis in hematological patients before and after allogeneic hematopoietic stem cell transplantation: implication for daily clinical practice. Eye (Lond). 2017 Oct;31(10):1417-1426. Karwacka E et all Pemphigoid-like ocular lesions in patients with graftversus-host disease following allogeneic bone marrow transplantation. Transplant Proc. 2006 Jan-Feb;38(1):292-4. | 50 patients or 53% were diagnosed as dry eye sufferers prior to HSCT. The incidence increased 77% or 72 patients post HSCT. Significant changes post HSCT: OSDI, TFBUT, MGD score, conjunctival injection; not so much Schirmer's. Pemphigoid-like ocular lesions in addition to keratitis sicca were seen in patients with graft-versus-host disease. |
| Kim S et al. Changes of meibomian glands in the early stage of post hematopoietic stem cell transplantation. Exp Eye Res. 2017 Oct;163:85-90. | "A significant increase was seen in the upper eyelid post-<br>HSCT meiboscore at 2 months and 3 months, and in the<br>total eyelid meiboscore at 3 months. |
| Kim SK 2006 Update on ocular graft versus host disease. Curr Opin Ophthalmol. 2006 Aug;17(4):344-8. | "Ocular graft versus host disease is a common sequela of allogeneic hematopoietic transplantation affecting up to 80% of chronic graft versus host disease patients. Clinical features of ocular graft versus host disease encompass all parts of the eye, from the lid to the choroids, although ocular graft versus host disease is most commonly viewed as a disease of the ocular surface, with the conjunctiva and lacrimal gland most commonly affected." |

| Reference | Ocular Changes Chronic GvHD |
|---|---|
| Kusne Y et al | "Clinical CSEF [conjunctival subepithelial fibrosis) may be |
| Conjunctival subepithelial fibrosis and meibomian gland | an important sign of GVHD impact on the ocular surface |
| atrophy in ocular graft-versus-host disease. Ocul Surf. | and may be relevant in oGVHD severity assessment." |
| 2017 Oct;15(4):784-788. | |
| Lin X, Cavanagh HD | "The most common presentations were |
| Ocular manifestations of graft-versus-host disease: 10 | keratoconjunctivitis sicca, cataract, blepharitis, ocular |
| years' experience. Clin Ophthalmol. 2015 Jul 3;9:1209-13. | hypertension, and filamentary keratitis. Visual acuity at |
| | presentation was 20/49; at the worst point in the disease was 20/115; and at most recent visit was 20/63.""they |
| | are prone to serious ocular complications such as corneal |
| | perforation and endophthalmitis." |
| Nassar A et al. | "Eyelid changes may occur in GVHD leading to |
| Ocular manifestations of graft-versus-host disease. Saudi | scleroderma-like changes. Patients may develop poliosis, |
| J Ophthalmol. 2013 Jul;27(3):215-22. | madarosis, vitiligo, lagophthalmos, and entropion. The |
| | cornea may show filamentary keratitis, superficial |
| | punctate keratitis, corneal ulcers, and peripheral corneal |
| | melting which may lead to perforation in severe cases. |
| | Scleritis may also occur which can be anterior or |
| | posterior. Keratoconjunctivis sicca appears to be the most |
| | common presentation of GVHD. The lacrimal glands may |
| | be involved with mononuclear cell infiltration of both the |
| | major and accessory lacrimal glands and decrease in tear production. Severe dry eye syndrome in patients with |
| | GVHD may develop conjunctival scarring, keratinization, |
| | and cicatrization of the conjunctiva." |
| Ogawa Y et al. | Ocular complications were listed for "chronic phase" |
| Dry eye as a major complication associated with chronic | Dry eye |
| graft-versus-host disease after hematopoietic stem cell | Meibomian gland dysfunction |
| transplantation. Cornea. 2003 Oct;22(7 Suppl):S19-27. | Retinal hemorrhage |
| | Aseptic conjunctivitis |
| | Lagophthalmos [inability to close eyelids completely] |
| | Corneal thinning |
| | Corneal melting |
| | Nasolacrimal obstruction |
| | Calcerous corneal degeneration Iritis |
| | Optic disc edema |
| | Cotton wool spots [fluffy white patches on retina] |
| | Cataract |
| Ogawa, Y. Sjögren's Syndrome, Non-Sjögren's Syndrome, | "In most cases [of chronic ocular GvHD] severe dry eye |
| and Graft-Versus-Host Disease Related Dry Eye. Invest. | progresses rapidly after the onset of symptoms and can |
| Ophthalmol. Vis. Sci. 2018;59(14):DES71-DES79. | lead to blindness. Despite improvements in the therapy |
| | for acute GVHD, specific therapies remain a substantial |
| | problem with little progressGlaucoma, cataract, |
| | infection, and corneal perforation should be prevented as |
| | side effects that occur after topical or systemic |
| | corticosteroid administration for preventing or treating |
| | GVHDThe 2014 NIH diagnostic criteria stated ocular cGVHD as a new onset of dry eye in the post-transplant |
| | patient. Additional symptoms may include photophobia, |
| | periorbital hyperpigmentation, or blepharitis. |
| | periorbital hyperpignientation, or biepharitis. |

| Reference | Ocular Changes Chronic GvHD |
|---|---|
| | Examination by ophthalmologists is necessary for diagnostic confirmation of keratoconjunctivitis sicca, cicatricial conjunctivitis, or punctate keratopathy. |
| | Schirmer's test was removed from the 2014 NIH diagnostic criteria." |
| Qiu Y et al. Manifestation of clinical categories of ocular graft-versushost disease. J Ophthalmol. 2018 Aug 8;2018:6430953. | Acute ocular GVHD predicts chronic ocular GVHD, is typified by acute conjunctivitis, increased mucus eye secretions, red eye, and lacrimation. Chronic ocular GVHD signs beyond severe eye include corneal lesions such as filamentary keratitis, corneal ulcer, and corneal vascularization, pseudomembrane formation, corneal epithelium loss. |
| Saboo US et al. Vision-Related Quality of Life in Patients with Ocular Graft-versus-Host Disease. Ophthalmology. 2015 Aug;122(8):1669-74. | "Compared with healthy subjects, patients with ocular GVHD reported reduced scores on all NEI-VFQ-25 subscales (each P < 0.001) with the exception of color vision (P = 0.11)." "Patients with ocular GVHD experience measurable impairment of vision-related QOL." |
| Shikari H et al. Onset of ocular graft-versus-host disease symptoms after allogeneic hematopoietic stem cell transplantation. Cornea. 2015 Mar;34(3):243-7. | Schirmer score can be "unreliable". Proposed reliance on incorporation of ophthalmological examination in BMT patients. |
| Shikari H et al. Ocular graft-versus-host disease: a review. Surv Ophthalmol. 2013 May-Jun;58(3):233-51. | Offers grading in acute and chronic GVHD. TABLE 1 Conjunctival Grading in Acute and Chronic GVHD Classification of Conjunctivitis in Acute GVHD <sup>66</sup> 0. None 1. Hyperemia 2. Hyperemia 3. Pseudomembranous conjunctivitis 4. Pseudomembranous conjunctivitis 4. Pseudomembranous conjunctivitis with corneal epithelial sloughing Classification of Conjunctivitis in Chronic GVHD <sup>135</sup> 0. None 1. Hyperemia 2. Palpebral conjunctival fibrovascular changes with or without epithelial sloughing 3. Palpebral conjunctival fibrovascular changes involving 25–75% of total surface area 4. Involvement of > 75% of total surface area with or without cicatricial entropion "Cicatricial conjunctival changes (Table 1) and superior limbic keratoconjunctivitis are commonly seen in chronic ocular GVHD. There is associated palpebral and fornicial conjunctival symblepharon with consequent lid scarring and disturbed lid anatomy (ectropion, entropion, meibomian gland atrophy, and punctal stenosis) Secondary epithelial changes such as punctate keratopathy develop with the formation of corneal filaments and painful erosions with resultant secondary infections, non-healing ulcerations, and corneal perforations." "KCS has been observed in 6977% of patients with chronic systemic GVHD and is an early sign of systemic involvement in extensive chronic GVHD." |
| Siebelmann S et al. | "Potential complications include visual loss, pain and damage to the ocular structures with, e.g. corneal |

| Reference | Ocular Changes Chronic GvHD |
|---|---|
| [Non-Invasive Diagnosis of Ocular Graft-versus-Host Disease]. Klin Monbl Augenheilkd. 2015 May;232(5):652-7. | ulcerations Available tests are mostly evaluated for usage in dry eye diagnosis but are, however, mostly unspecific for diagnosing ocular GvHD reliably." |
| Sun YC et al. Impact of Ocular Chronic Graft-versus-Host Disease on Quality of Life. Biol Blood Marrow Transplant. 2015 Sep;21(9):1687-91. | "Of the 284 chronic GVHD patients, 116 (41%) had ocular GVHD within 3 months of chronic GVHD diagnosis ("early ocular GVHD"). Late ocular GVHD (new onset > 3 months after chronic GVHD diagnosis) occurred in 64 patients. Overall cumulative incidence at 2 years was 57%." |
| Tung Cl<br>Graft versus host disease: what should the oculoplastic<br>surgeon know? Curr Opin Ophthalmol. 2017 Sep;<br>28(5):499-504. | "Ocular GVHD occurs as a common immune-mediated complication of hematopoietic stem cell transplantation that presents as a Stevens-Johnson-like syndrome in the acute phase or a Sjögren-like syndrome in the chronic phase. Cicatricial conjunctivitis may be underreported in ocular GVHD. The spectrum of oculoplastic manifestations includes GVHD of the skin, cicatricial entropion, nasolacrimal duct obstruction, and lacrimal gland dysfunction. Surgical treatment is indicated for patients with significant corneal complications from entropion. Surgical approach to repair of nasolacrimal duct obstruction is presented in this review, including modified approaches for treating patients at risk for keratitis sicca." |
| Westeneng AC et al Ocular graft-versus-host disease after allogeneic stem cell transplantation. Cornea. 2010 Jul;29(7):758-63. | "Over time, ocular GvHD developed in 54% of patients and consisted mainly of dry eyes and conjunctivitis, which increased in severity during follow-up; blepharitis and uveitis were less often encounteredeye symptoms affecting activities of daily living were reported in 24 of 54 patients (44%) and 16 of 54 patients (30%) experienced temporary loss of visual acuity of more than 2 Snellen lines, only 1 developed permanent unilateral loss (counting fingers) because of ischemic vasculopathy." |

## **APPENDICES**

## SCHEDULE OF VISITS AND ASSESSMENTS

## Visits 1-7

| Blue = Conducted at DFCI | | Study Treatment Phase | | | Placebo Cross-over Phase | | | |
|---|---|---|---|---|---|---|---|---|
| Black = Conducted at MEEI | Visit 1<br>(Screening) | Visit 2 Baseline &<br>First Drug Application | | Visit 3 | Visit 3 Visit 4 Visit 5 | | Visit 6 | Visit 7 |
| | Day -14 to -1 | Day 1 | Day 1 | Day 14±2 | Day 42±3 | Day 70±3 | 3 weeks | 6 weeks |
| Procedure | | Pre-Dose | 30-60 min<br>Post-Dose | | | | | |
| 2-digit screening number | X | | | | | | | |
| Informed consent | X | | | | | | | |
| Visual acuity (current correction) | X | | | | | X | | |
| NIH Ocular GvHD Score | X | | | | | X | | X <sup>2</sup> |
| Facial photo | | X | | | | X | | X |
| Slit lamp biomicroscopy | X | | | X | X | X | X | X |
| Undilated fundoscopy exam | X | | | | | X | | |
| Corneal and conjunctival staining | X | | | X | X | X | X | X |
| Intraocular pressure | X | | | | | X | | X |
| Inclusion/Exclusion criteria | X | | | | | | | |
| Medical/Ophthalmology history and updates | X | X | | X | X | X | X | X |
| Prior and concomitant medication query | X | X | | X | X | X | X | X |
| Concomitant medications (BMT) | X | | | | X | X | | X |
| Medical history & physical (BMT) | X | | | | | | | |
| Demographic data | X | | | | | | | |
| Video of face & eyes (1 minute) | | X | X | X | X | X | X | X |
| TearScan examination | | X | X | X | X | X | X | X |
| Urine pregnancy test | X | | | | | X | | |
| Modified SANDE questionnaire | X | | | X | X | X | X | X |
| GLIA Ocular Surface Disease Symptoms<br>Questionnaire | X | X | X | X | X | X | X | X |
| Adverse event query | | | X | X | X | X | X | X |
| Screen Pass/Fail | X | | | | | | | |
| 3-digit random number | X | | | | | | | |
| BMT systemic evaluation & GvHD assessment | X | | | | X | X | | X |
| Standard GvHD, CBC, and metabolic labs | X | | | | X | X | | X |
| Endocrine panel | X | | | | X | X | | X |
| Daily diary and ocular medication log collected | | | | X | X | X | X | X |
| Study drug collected/ accountability | | | | X | X | X | X | X |
| Study drug application (in-clinic) | | X | | | | | | |
| Study drug dispensed | | X | | X | X | X | X | |
| Daily diary & ocular medication log dispensed | | | X | X | X | X | X | |

<sup>&</sup>lt;sup>2</sup> Added as protocol deviation to original protocol v4.

# SCHEDULE OF VISITS AND ASSESSMENTS Visits 8-9 Long Term Open Label

| Blue = Conducted at DFCI | Visit 8 | Visit 9 |
|---|---|---|
| Black = Conducted at MEEI | 66 ± 6 weeks<br>(15 months) | 117 ± 6 weeks<br>(27 months) |
| Procedure | | |
| Informed consent for long term open phase | X | X |
| Visual acuity (current correction) | X | X |
| NIH Ocular GvHD Score | X | X |
| Facial photo | X | X |
| Slit lamp biomicroscopy | X | X |
| Undilated fundoscopy exam | X | X |
| Corneal and conjunctival staining | X | X |
| Intraocular pressure | X | X |
| Ophthalmology updates | X | X |
| Concomitant medications (BMT) | X | X |
| Video of face & eyes (1 minute) | X | X |
| TearScan examination | X | X |
| Urine pregnancy test | X | X |
| Modified SANDE questionnaire | X | X |
| GLIA Ocular Surface Disease Symptoms Questionnaire | X | X |
| Adverse event query | X | X |
| BMT systemic evaluation & GvHD assessment | X | X |
| Standard GvHD, CBC, and metabolic labs | X | X |
| Endocrine panel | X | X |

| Initials | :: Subject #: | Date: | Examiner: | |
|---|---|---|---|---|
| | Symptom A | Assessment iN Dry I | Eye (SANDE) Question | naire |
| | E COMPLETE THE FOLLO<br>UR DRY EYE SYMPTOMS | | REGARDING THE FREQU | JENCY AND SEVERITY |
| 1. <u>Fre</u> | quency of symptoms: | | | |
| Please<br>irritat | e place an 'X' on the line ed: | to indicate <u>how oft</u> o | <u>en</u> , on average, your ey | res feel <b>dry and/or</b> |
| Left | Rarely | | | _ All the time |
| Right | Rarely | | | _ All the time |
| 2. <u>Sev</u> | erity of symptoms: | | | |
| | e place an 'X' on the line ss and/or irritation: | to indicate <u>how sev</u> | <u>ere</u> , on average, you fe | el your symptoms of |
| Left | Very Mild | | | Very Severe |
| Right | Very Mild | | | Very Severe |

| | | | | Sportsor, GLIA LL |
|---|---|---|---|---|
| GLIA™ OCULAR SURF | ACE DISEASE SYMPTOMS QU | ESTIONNAIRE - CLINIC RECO | ORD | |
| Initials: Subject #: | Date: | Examiner: | - | |
| Grade by placing X on the | line from 'None' to 'Most severe' | None Most | | |
| | Baseline Time | <b>::</b> | Post-application 30-90 mir | 1 Time: |
| | OD | os | OD | os |
| Ocular discomfort | None Most | None Most | None Most | None Most |
| Dryness | None Most | None Most | None Most | None Most |
| Grittiness | None Most | None Most | None Most | None Most |
| Burning | None Most | None Most | None Most | None Most |
| Stinging | None Most | None Most | None Most | None Most |
| Foreign body sensation | None Most | None Most | None Most | None Most |
| Ocular pain | None Most | None Most | None Most | None Most |
| Conjunctival redness | None Most | None Most | None Most | None Most |
| Additional notes below: | Datails and other acular symptoms) | | ı | |

Additional notes below: (Details and other ocular symptoms)

| | | | | Sponsor: GLIA LI |
|---|---|---|---|---|
| GLIA™ OCULAR SURF. | ACE DISEASE SYMPTOMS QU | ESTIONNAIRE - CLINIC RECO | ORD | |
| Initials: Subject #: _ | Date: | Examiner: | - | |
| Grade by placing X on the l | ine from 'None' to 'Most severe' | None Most | ] | |
| | Baseline Time | e: | Post-application 30-90 min | 1 Time: |
| | OD | os | OD | os |
| Itching | None Most | None Most | None Most | None Most |
| Mucus discharge | None Most | None Most | None Most | None Most |
| Photophobia | None Most | None Most | None Most | None Most |
| Blurred or cloudy vision | None Most | None Most | None Most | None Most |
| Airflow sensitivity | None Most | None Most | None Most | None Most |
| Lid redness | None Most | None Most | None Most | None Most |
| Lid sticking | None Most | None Most | None Most | None Most |
| | | | , | , |

Additional notes below: (Details and other ocular symptoms)

## Ocular GvHD Evaluations & Scoring in clinic

| Evaluation | Method | Scoring |
|---|---|---|
| Pre-fluorescein stain | | |
| Visual acuity | Eye chart, OD and OS | See below |
| Slit lamp: | Visual or slit lamp | |
| <u>Lids</u> : Lid margin erythema, | | None Most severe |
| edema, ulceration, notches, | | |
| entropion/ ectropion, | | None Most severe |
| trichiasis/madarosis, floppy | | |
| eyelids, hordeolum; | | |
| Conjunctiva: Hyperemia, | | |
| cicatricial changes, | | |
| pseudomembranes, chalasis; | | |
| Cornea: Edema, ulcers, | | |
| filamentous keratitis, thinning, | | |
| corneal neovascularization, | | |
| scars, conjunctivial epithelium | | |
| invasion, limbal thickening; | | |
| Anterior chamber: Cells, flare; | | |
| <u>Lens opacity</u> | | |
| Tear film evaluation + lid | TearScan | 0,1, 2, 3 |
| margin | | |
| After fluorescein stain | | |
| Fluorescein staining | Slit lamp | None Most severe |
| | | None Most severe |
| | | MOST Severe |
| Intraocular pressure | Applanation tonemetry | Reading in mm Hg |

## **NIH Ocular GvHD Score**

| SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|
| No symptoms | Mild dry eye symptoms not affecting ADL (requirement of lubricant eye drops ≤ 3 x per day) | Moderate dry eye symptoms partially affecting ADL (requiring lubricant eye drops > 3 x per day or punctal plugs), WITHOUT new vision impairment due to KCS | Severe dry eye symptoms significantly affecting ADL (special eyeware to relieve pain) OR unable to work because of ocular symptoms OR loss of vision due to KCS |

## Tearscan™ Examinations

The TearScan enables non-invasive viewing of the lipid film on the surface of the eye that does not require the use of fluorescein staining. It provides a white light source that encircles the eye, to allow illumination of the ocular surface. A video camera inserted in the center of the ring of light, and connected to a computer, allows viewing and video recording of the tear film

During the examination, a one-minute video that includes 3 natural blinks should be recorded.

| The | grading | will | he | from | 0 | to | 3. |
|------|---------|--------|----------|--------|---|---------------|----|
| 1110 | graumg | VV 111 | $\sigma$ | 110111 | v | $\iota \circ$ | J. |

- 0 = no discernible tear film
- 1 = thin tear film
- 2 = moderate tear film
- 3 = copious tear film

| Initials: | Subject #: | Date: | Examiner: |
|-------------|-------------|-------|-----------|
| OD (right | eye) Score: | | |
| OS (left ey | e) Score: | | |
| Pod ovo lid | I. Vos N | 0 | |



## **Visual Acuity**

Distance and near Snellen acuity in current glasses if wearing, (or no glasses if not wearing), then pinhole.

| OD (right eye) |
|----------------|
| OS (left eve) |

## SLIT LAMP BIOMICROSCOPY WITHOUT STAINING - OCULAR GVHD

| Initials: | Subject #: | Date | e: | | Examiner: | | |
|---|---|---|---|---|---|---|---|
| Indicate a Grade by placing X on the line for all POSITIVE FINDINGS: | | | | | | | |
| If finding present, Chec | k NCS or CS (NC | S = Non Clini | cally Sig | gnificant | CS = Clinical | lly Significant) | |
| Lids<br>☐ No positive findings | | OD | | | | os | |
| Erythema | None | Most severe | □cs | □ncs | None | Most severe | □cs □ncs |
| Edema | None | Most severe | □cs | □ncs | None | Most severe | □cs □ncs |
| Lid margin ulceration | None | Most severe | □cs | □ncs | None | Most severe | □cs □ncs |
| Lid margin notches | None | Most severe | □cs | □ncs | None | Most severe | □cs □ncs |
| Entropion/Ectropion | None | Most severe | □cs | □ncs | None | Most severe | □cs □ncs |
| Trichiasis/Madarosis | None | Most severe | □cs | □ncs | None | Most severe | □cs □ncs |
| Floppy eyelids | None | Most severe | □cs | □ncs | None | Most severe | □cs □ncs |
| Hordeolum (stye) | None | Most severe | □cs | □ncs | None | Most severe | □cs □ncs |
| Other pathology, specify: | : | | | | | | |
| | _□cs □ncs;_ | | | □cs | □NCS; | | _□cs □ncs |
| Conjunctiva ☐ No positive findings | | | | | | 000 | |
| | | OD | | | | OS | |
| Hyperemia | None | Most severe | □cs | □ncs | None | Most severe | □cs □ncs |
| Hyperemia Cicatricial changes | None | | | □ncs | None | | □cs □ncs |
| | | Most severe | □cs | | | Most severe | |
| Cicatricial changes | None | Most severe | □cs<br>□cs | □ncs | None | Most severe | □cs □ncs |
| Cicatricial changes Pseudomembranes | None None None | Most severe Most severe | □cs<br>□cs | □ncs | None | Most severe Most severe | □cs □ncs □cs □ncs |
| Cicatricial changes Pseudomembranes Chalasis | None None None | Most severe Most severe Most severe | □cs<br>□cs | □ncs □ncs □ncs | None | Most severe Most severe | □cs □ncs □cs □ncs |
| Cicatricial changes Pseudomembranes Chalasis | None None | Most severe Most severe Most severe | □cs<br>□cs | □ncs □ncs □ncs | None None | Most severe Most severe | □cs □ncs □cs □ncs □cs □ncs |
| Cicatricial changes Pseudomembranes Chalasis Other pathology, specify: | None None | Most severe Most severe Most severe | □cs<br>□cs<br>□cs | □ncs □ncs □ncs | None None | Most severe Most severe Most severe | □cs □ncs □cs □ncs □cs □ncs |
| Cicatricial changes Pseudomembranes Chalasis Other pathology, specify: Cornea No positive findings | None None CS NCS; | Most severe Most severe Most severe | □cs □cs □cs | □NCS □NCS □NCS | None None None | Most severe Most severe Most severe | □cs □ncs □cs □ncs □cs □ncs □cs □ncs |

| Indicate a Grade by placing X on the line for all POSITIVE FINDINGS: | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| If finding present, Chec | k NCS or CS (NCS | s = Non Clini | cally S | ignifican | t CS = Clinicall | y Significant) | | |
| Corneal thinning | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Corneal neovascularization | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Scars | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Conjunctival epithelium invasion | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Limbal thickening | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Other pathology, specify: | | | 1 | | | | | |
| | _□cs □ncs; _ | | | | S □NCS; | | □cs | □NCS |
| Anterior Chamber ☐ No positive findings | | OD | | | | os | | |
| Cells | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Flare | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Other pathology, specify: | | | | | | | • | |
| | _□cs □ncs; _ | | | | S □NCS; | | _□cs | □NCS |
| <u>Lens Status</u> | OD | | | | OS | | | |
| | □Phakic | | | | □Phakic | | | |
| | □Pseudopha | kic | | | □Pseudophakid | ; | | |
| | □Aphakic | | | | □Aphakic | | | |
| Lens Opacity<br>(Phakic Eye ONLY)<br>□ No positive findings | OD | | | | os | | | |
| | □ <sub>0</sub> □+1□+ <sub>2</sub> □ | +3 | □cs | □ncs | $\square_0\square$ +1 $\square$ +2 $\square$ +3 | | □cs | □ncs |
| Comments: | | | | | | | | |

#### **FLUORESCEIN STAINING**

| | Initials: | _ Subject #: | Date: | Examiner: | <del></del> |
|---|---|---|---|---|---|
| Sodiun | n Fluorescein stri | ips (thin tipped, DET | TTM strips preferre | d) should be moisten | ed with one or two drops of |
| sterile | irrigating or salin | ne solution. Apply r | noistened tip to c | onjunctiva or fornix. | The subject should blink |
| several | l times after appli | ication and wait for 2 | 2 minutes before 6 | examination. | |

| Indicate a Grade by placing X on the line for all POSITIVE FINDINGS: | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| If finding present, Ched | ck NCS or CS (N | CS = Non Clin | ically S | Significant | CS = Clir | nically Significant) | | |
| Cornea ( C) ☐ No positive findings | | OD | | | | os | | |
| Inferior | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Superior | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Central | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Other pathology, specify | | | | □cs | i □ncs; | | _□cs | □ncs |
| Conjunctiva ☐ No positive findings | | OD | | | | os | | |
| Inferior | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Superior | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Temporal | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Nasal | None | Most severe | □cs | □ncs | None | Most severe | □cs | □ncs |
| Other pathology, specify | : | | | | | | | |
| | _□cs □ncs; | | | □cs | □ NCS; | | _□cs | □ncs |



## **UNDILATED FUNDOSCOPY - OCULAR GVHD**

(To be performed only at Screening and Last Visit)

Initials: \_\_\_\_\_ Subject #:\_\_\_\_ Date: \_\_\_\_ Examiner: \_\_\_\_\_

| | Check Normal or Abnormal | | OD | | | | | os | |
|---|---|---|---|---|---|---|---|---|---|
| (If Abnormal, check NCS)* | CS or | Normal | mal Abnormal | | Abnormal | Normal | mal Abnormal | | Abnormal |
| NC3) | | | NCS | CS | comments | | NCS | CS | comments |
| Vitreous | | | | | | | | | |
| Optic nerve | | | | | | | | | |
| Macula | | | | | | | | | |
| Vessels | | | | | | | | | |
| Cup to disc ratio | | | | | | | | | |
| Jrine Test Strip: HCG One Step Pregnancy Test or similar. Jrine Collection: A nurse will dispense a urine collection cup for urine collection. | | | | | | | | | |
| Test Procedure: | <b>Procedure:</b> Follow directions, but usually the test strip is dipped into the urine for 3 seconds, and laid flat for reading within 5 minutes. | | | | | | | | |
| Initials: Subje | ect #: | Date: | | | _ Examiner: | | | _ | |

| CBC and DIFFERENTIAL | Normal Range |
|----------------------|------------------|
| WBC | 3.81 - 8.94 K/uL |
| RBC | 4.35 - 5.61 M/uL |
| HGB | 12.5 - 16.3 g/dL |
| HCT | 37.1 - 49.5 % |
| PLT | 152 - 440 K/uL |
| MCV | 79.0 - 97.0 fL |
| MCH | 26.2 - 32.0 pg |
| MCHC | 33.3 - 35.7 g/dL |
| RDW | 12.1 - 16.0 % |
| MPV | 7.0 - 10.8 fl |
| NRBC | 0.00 /100 WBCs |
| ABSOLUTE NRBC | K/uL |
| NEUTS | 46.5 - 82.4 % |
| EOSINOPHIL | 0.1 - 6.0 % |
| BASOPHIL | 0.1 - 1.1 % |
| LYMPHS | 8.5 - 32.7 % |
| MONOS | 5.4 - 14.2 % |
| ABSOLUTE NEUTS | 2.23 - 6.11 K/uL |
| ABSOLUTE EOS | 0.00 - 0.52 K/uL |
| ABSOLUTE BASO | 0.00 - 0.11 K/uL |
| ABSOLUTE LYMPHS | 0.21 - 2.74 K/uL |
| ABSOLUTE MONOS | 0.2 - 0.87 K/uL |

| COMPREHENSIVE METABOLIC PANEL | Normal Range |
|-------------------------------|-------------------|
| SODIUM | 135 - 145 mmol/L |
| POTASSIUM | 3.5 - 5.0 mmol/L |
| CHLORIDE | 98 - 108 mmol/L |
| CO2 | 23 - 32 mmol/L |
| BUN | 9 - 25 mg/dL |
| CREATININE | 0.7 - 1.3 mg/dL |
| GLUCOSE | 70 - 100 mg/dL |
| ALBUMIN | 3.7 - 5.4 g/dL |
| TOTAL PROTEIN | 6.0 - 8.0 g/dL |
| CALCIUM | 8.8 - 10.5 mg/dL |
| ALKALINE PHOSPHATASE | 36 - 118 U/L |
| TOTAL BILIRUBIN | 0.2 - 1.2 mg/dL |
| AST | 9 - 30 U/L |
| ALT | 7 - 52 U/L |
| GLOBULIN | 2.3 - 4.2 g/dL |
| EGFR | >59 mL/min/1.73m2 |
| ANION GAP | 5 - 17 mmol/L |

| OTHER STANDARD GVHD | Normal Range |
|---|---|
| TACROLIMUS | 3.0 - 15.0 ng/mL |
| VITAMIN D Total, 25-OH (D2 and D3)<br>Sunquest Lab, OHDT | 20-80 ng/mL |
| T4 (thyroxine), Total, Serum | 11 -19 years: 5.9-13.2 μg/dL<br>Adult (> or =20 years): 4.5-11.7 μg/dL |
| T4 (thyroxine), Free, Serum | 11-19 years: 1.0-1.6 ng/dL<br>Adult (> or =20 years): 0.9-1.7 ng/dL |
| T3 (triodothyronine), Total, Serum | 11-19 years: 91-218 ng/dL<br>Adult (> or =20 years): 80-200 ng/dL |
| ACTH (adrenocorticotropic hormone), Plasma | 7.2-63 pg/mL (a.m. draws) |
| TSH (thyroid stimulating hormone), Serum | 0.27 - 4.20 μIU/mL |

| ENDOCRINE PANEL | Normal Range |
|---|---|
| DHEA-S (dehydroepiandrosterone sulfate), | 18-30 years: 105-728 μg/dL |
| Serum | 31-40 years: 57-522 μg/dL |
| | 41-50 years: 34-395 μg/dL |
| | 51-60 years: 20-299 μg/dL |
| | 61-70 years: 12-227 μg/dL |
| | > or =71 years: 6.6-162 μg/dL |
| ESTRADIOL, Serum | Follicular Phase 27-156 pg/mL |
| | Mid Cycle Peak 48-314 pg/mL |
| | Luteal Phase 33-298 pg/mL |
| | Postmenopausal <50 pg/mL |
| FSH (follicle stimulating hormone), Serum | Male 1.6-8.0 mIU/mL |
| | Female |
| | Follicular Phase 2.5-10.2 mIU/mL |
| | Mid-Cycle Peak 3.1-17.7 mIU/mL |
| | Luteal Phase 1.5- 9.1 mIU/mL |
| | Postmenopausal 23.0-116.3 mIU/mL |
| LH (luteinizing hormone), Serum | Male |
| | 18-59 Years 1.5-9.3 mIU/mL |
| | ≥60 Years 1.6-15.2 mIU/mL |
| | Female |
| | Follicular Phase 1.9-12.5 mIU/mL |
| | Mid-Cycle Peak 8.7-76.3 mIU/mL |
| | Luteal Phase 0.5-16.9 mIU/mL |
| | Postmenopausal 10.0-54.7 mIU/mL |
| PTH (Parathyroid Hormone), Serum | 15-65 pg/mL |
| PROGESTERONE, Serum | MALES > or =18 year: <0.20 ng/mL |
| | FEMALES > or =18 years: |
| | -Follicular phase: < or =0.89 ng/mL |
| | -Ovulation: < or =12 ng/mL |
| | -Luteal phase: 1.8-24 ng/mL |
| | -Post-menopausal: < or =0.20 ng/mL |
| | -Pregnancy |
| | - 1st trimester: 11-44 ng/mL |
| | - 2nd trimester: 25-83 ng/mL |

| ENDOCRINE PANEL | Normal Range |
|---|---|
| ENDOCKINE I ANEE | - 3rd trimester: 58-214 ng/mL |
| | - 3rd trimester: 38-214 rig/file |
| TESTOSTERONE, Total and Free, Serum | TESTOSTERONE, FREE |
| Mayo Clinic test code TGRP | Males (adult): |
| , | 20-<25 years: 5.25-20.7 ng/dL |
| | 25-<30 years: 5.05-19.8 ng/dL |
| | 30-<35 years: 4.85-19.0 ng/dL |
| | 35-<40 years: 4.65-18.1 ng/dL |
| | 40-<45 years: 4.46-17.1 ng/dL |
| | 45-<50 years: 4.26-16.4 ng/dL |
| | 50-<55 years: 4.06-15.6 ng/dL |
| | 55-<60 years: 3.87-14.7 ng/dL |
| | 60-<65 years: 3.67-13.9 ng/dL |
| | 65-<70 years: 3.47-13.0 ng/dL |
| | 70-<75 years: 3.28-12.2 ng/dL |
| | 75-<80 years: 3.08-11.3 ng/dL |
| | 80-<85 years: 2.88-10.5 ng/dL |
| | 85-<90 years: 2.69-9.61 ng/dL |
| | 90-<95 years: 2.49-8.76 ng/dL |
| | 95-100+ years: 2.29-7.91 ng/dL |
| | Females (adult): |
| | 20-<25 years: 0.06-1.08 ng/dL |
| | 25-<30 years: 0.06-1.06 ng/dL |
| | 30-<35 years: 0.06-1.03 ng/dL |
| | 35-<40 years: 0.06-1.00 ng/dL |
| | 40-<45 years: 0.06-0.98 ng/dL |
| | 45-<50 years: 0.06-0.95 ng/dL |
| | 50-<55 years: 0.06-0.92 ng/dL |
| | 55-<60 years: 0.06-0.90 ng/dL |
| | 60-<65 years: 0.06-0.87 ng/dL |
| | 65-<70 years: 0.06-0.84 ng/dL |
| | 70-<75 years: 0.06-0.82 ng/dL |
| | 75-<80 years: 0.06-0.79 ng/dL |
| | 80-<85 years: 0.06-0.76 ng/dL |
| | 85-<90 years: 0.06-0.73 ng/dL |
| | 90-<95 years: 0.06-0.71 ng/dL |
| | 95-100+ years: 0.06-0.68 ng/dL |
| | TESTOSTERONE, TOTAL |
| | Males |
| | 17-18 years: 300-1,200 ng/dL |
| | • |
| | > or =19 years: 240-950 ng/dL<br>Females |
| | 17-18 years: 20-75 ng/dL |
| | > or =19 years: 8-60 ng/dL |

| ا ما مانا | Cub | inat # |
|-----------|-----|---------|
| nitials: | Sub | ject #: |

## Home Record of Actual Ocular Medication and Artificial Tear Use

(Record date and number of times used per day and night)

| | GV-1 | Ocular Med 1 | Ocular Med 2 | Artificial<br>Tears & Gels | Artificial<br>Tears & Gels | Ocular Med 4 | Ocular Med 5 | Ocular Med 6 |
|---|---|---|---|---|---|---|---|---|
| | | | | Use only when necessary | | | | |
| Name of medication | | | | | | | | |
| Date | | | | | | | | |

| DATE: | DAY OF WEEK | : | | |
|---|---|---|---|---|
| Initials: Subje | ect #: Rev | iewed by / date: _ | | |
| Grade by placing X or | n the line from 'None' to 'I | Most severe' | None | Most |
| Baseline Time: | | | | |
| | Ol | D | ( | os |
| Ocular discomfort | None | Most | None | Most |
| Dryness | None | Most | None | Most |
| Grittiness | None | Most | None | Most |
| Burning | None | Most | None | Most |
| Stinging | None | Most | None | Most |
| Foreign body sensation | None | Most | None | Most |
| Ocular pain | None | Most | None | Most |
| Conjunctival redness | None | Most | None | Most |
| Itching | None | Most | None | Most |
| Mucus discharge | None | Most | None | Most |
| Photophobia | None | Most | None | Most |
| Blurred or cloudy vision | None | Most | None | Most |
| Airflow sensitivity | None | Most | None | Most |
| Lid redness | None | Most | None | Most |
| Lid sticking | None | Most | None | Most |
| Additional notes bel | ow: (Details and other oc | ular symptoms) | | |

| Pro | o-Ocular 1% | Topical Gel |
|-----|-------------|-------------|
| | Snonsc | r: GHA HC |

| | 0 1: |
|-----------|------------|
| Initials: | Subject #: |

## **ADVERSE EVENT LOG**

| Visit<br>Number | Report date<br>(mm/dd/yyyy) | Adverse event | Relationship<br>to study<br>drug(1, 2, or 3) | Adverse event onset date (mm/dd/yyyy) | Adverse event<br>end date<br>(mm/dd/yyyy) | Severity<br>(1, 2,or 3) | Action taken with study drug(1-, 2, 3, or 4) | Specify, if<br>action taken<br>with study<br>drug="4. Other" | Outcome<br>(1, 2,or 3) | Serious<br>adverse<br>event<br>(Yes/No) |
|---|---|---|---|---|---|---|---|---|---|---|

## Enter numerical responses for following Questionnaire categories

Action taken with study drug: Relationship to study drug: Outcome: Severity: 1. None 1. None 1. Resolved 1. Mild 2. Possibly related 2. Permanently Discontinued\* 2. Ongoing 2. Moderate 3. Probably related 3. Temporarily Discontinued 3. Lost to follow-up 3. Severe

4. Other(specify)

<sup>\*</sup> Complete study discontinuation form